CLINICAL TRIAL: NCT02820805
Title: The Effect of Dietary Carbohydrate Consumption on Memory Performance and Mood in Normal Weight and Overweight/Obese Children
Brief Title: Dietary Carbohydrate Consumption on Memory Performance and Mood in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, School of Nutrition, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB2016-060
Record Dates: First submitted 2016-06-27; First posted 2016-07-01 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Cognitive Ability, General
Keywords: children; dietary carbohydrates; solanum tuberosum; cognition; memory; emotions; blood glucose
MeSH Terms: interventions — lunatusin, Phaseolus lunatus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Meal skipping (Experimental): No meal given
  Interventions: Other: Meal Skipping
- Mashed potatoes (Experimental): Carbohydrate Test Meal (50 g of available carbohydrates)
  Interventions: Other: Mashed potatoes
- French fries (Experimental): Carbohydrate Test Meal (50 g of available carbohydrates)
  Interventions: Other: French fries
- Hash browns (Experimental): Carbohydrate Test Meal (50 g of available carbohydrates)
  Interventions: Other: Hash browns
- Rice (Experimental): Carbohydrate Test Meal (50 g of available carbohydrates)
  Interventions: Other: Rice
- Beans (Experimental): Carbohydrate Test Meal (50 g of available carbohydrates)
  Interventions: Other: Beans

INTERVENTIONS:
Other: Meal Skipping — No meal
  Arms: Meal skipping
Other: French fries — 50g of available carbohydrates meal
  Arms: French fries
Other: Mashed potatoes — 50g of available carbohydrates meal
  Arms: Mashed potatoes
Other: Hash browns — 50g of available carbohydrates meal
  Arms: Hash browns
Other: Rice — 50g of available carbohydrates meal
  Arms: Rice
Other: Beans — 50g of available carbohydrates meal
  Arms: Beans

SUMMARY:
The purpose of this study is to determine the effect of carbohydrates on blood glucose levels, subjective appetite, mood, and memory performance in 9 to 14 year old normal weight (NW) and overweight or obese (OW/OB) children.

DETAILED DESCRIPTION:
NW and OW/OB children, 9-14 years of age, will participate in the experiment. The effect of 5 different meals (mashed potatoes, hash browns, French fries, rice, or beans matched by 50g of available carbohydrate) and meal skipping will be examined. On six separate mornings, one of the meals or no meal will be provided in a random order upon their arrival. Blood glucose, subjective appetite, and mood will be measured at baseline, 10, 30, 60, 120, and 180 minutes after meal consumption. Cognitive performance will be measured using an immediate and delayed word recall test, and two to three executive function tasks at 10, 30, 60, 120, and 180 minutes after meal consumption.

ELIGIBILITY:
Inclusion Criteria:

* be between 9 and 14 years of age
* be healthy, and have been born at term
* be a native English speaker
* not be taking any medications
* not have allergies to potatoes, rice, or beans.
* normal body weight (between the 5th and 85th BMI percentile for age and gender)
* OW/OB (>85th BMI percentile for age and gender)

Exclusion Criteria:

* Food sensitivities, allergies, or dietary restrictions
* Health, learning, emotional, or behaivoural problems
* Receiving any medications

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 10, 30, 60, 120, 180 minutes after meal consumption
  Participants will participate in a battery of tests that include two learning and memory tasks and two attention tasks at 10, 30, 60, 120, and 180 minutes after meal consumption.

SECONDARY OUTCOMES:
Blood glucose response | Baseline, 10, 30, 60, 120, and 180 minutes after meal consumption
  Blood will be collected at baseline, 10, 30, 60, 120, and 180 minutes after meal consumption to observe glycemic responses to 50g available carbohydrates from mashed potatoes, potato pancakes, French fries, rice, or beans
Subjective Appetite and Mood | Baseline, 10, 30, 60, 120, and 180 minutes after meal consumption
  Participants will complete subjective ratings on appetite (e.g., desire to eat, hunger, fullness) and mood (e.g. anger, happiness, excitement, sleepiness) at baseline, 10, 30, 60, 120, and 180 minutes after meal consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD., Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided